CLINICAL TRIAL: NCT01520753
Title: A Randomised, Double-blind, 4-week, Crossover Trial on Two Treatment Regimens With Biphasic Insulin Aspart 70 and 50 in Patients With Type 2 Diabetes
Brief Title: Comparison of Two Biphasic Insulin Aspart Treatments in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1074
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 70 (Experimental)
  Interventions: Drug: biphasic insulin aspart 70
- BIAsp 70 + BIAsp 50 (Experimental)
  Interventions: Drug: biphasic insulin aspart 70; Drug: biphasic insulin aspart 50

INTERVENTIONS:
Drug: biphasic insulin aspart 70 — Administered subcutaneously (s.c., under the skin) at breakfast, lunch and dinner
  Arms: BIAsp 70
Drug: biphasic insulin aspart 70 — Administered subcutaneously (s.c., under the skin) at breakfast and lunch
  Arms: BIAsp 70 + BIAsp 50
Drug: biphasic insulin aspart 50 — Administered subcutaneously (s.c., under the skin) at dinner
  Arms: BIAsp 70 + BIAsp 50

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two different active treatment regimens of biphasic insulin aspart in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Duration of diabetes for longer than 12 months
* Body mass index (BMI) below 35.0 kg/m^2
* HbA1c below 11.0 %
* Treatment with BHI (biphasic human insulin) 20 or 30 twice daily for at least three months and in the last month as sole anti-diabetic treatment (i.e., no additional oral hypoglycaemic medication or daily use of short-acting insulin supplement)

Exclusion Criteria:

* Current treatment with agents affecting glucose metabolism
* History of drug or alcohol dependence
* Impaired hepatic function
* Impaired renal function
* Cardiac disease
* Proliferative retinopathy
* Recurrent severe hypoglycaemia or advanced neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1999-03; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Fasting serum glucose

SECONDARY OUTCOMES:
24-hour serum glucose profiles
24-hour insulin profiles
Incidence of hypoglycaemic episodes
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Århus C, Denmark

REFERENCES:
- [Result] Ejskjaer N, Rasmussen M, Kamp N, Lindholm A, Christiansen JS. Comparison of thrice daily 'high' vs. 'medium' premixed insulin aspart with respect to evening and overnight glycaemic control in patients with type 2 diabetes. Diabetes Obes Metab. 2003 Nov;5(6):438-45. doi: 10.1046/j.1463-1326.2003.00299.x. PMID 14617230
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com